CLINICAL TRIAL: NCT06882811
Title: Clinical Study on Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Sepsis
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells Treatment in Sepsis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, xu xiang, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024404
Record Dates: First submitted 2025-03-17; First posted 2025-03-19 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 135 patients are infused with 1×10⁸ stem cells per session (Experimental)
  Interventions: Biological: CD83-positive MSC; Biological: regulatory MSC
- 45 patients are infused with equal volume of control solution (Sham Comparator)
  Interventions: Other: control solution

INTERVENTIONS:
Biological: CD83-positive MSC — 90 patients are infused with 1×10⁸ stem cells per session and receive regulatory treatment
  Arms: 135 patients are infused with 1×10⁸ stem cells per session
Biological: regulatory MSC — 45 patients are infused with 1×10⁸ stem cells per session and receive regulatory treatment
  Arms: 135 patients are infused with 1×10⁸ stem cells per session
Other: control solution — 45 patients are infused with equal volume of control solution and receive regulatory treatment
  Arms: 45 patients are infused with equal volume of control solution

SUMMARY:
The primary objective: To evaluate the efficacy of intravenous infusion of universal UC-MSCs and CD83+MSCs subpopulation injection in the treatment of sepsis by using the 28-day survival rate of the subjects as the primary efficacy criterion.The secondary objectives: 1. To systematically evaluate the safety of universal UC-MSCs and CD83+MSCs subpopulation in the treatment of sepsis; 2. To provide theoretical basis and clinical research data for establishing a safe, effective and feasible clinical treatment plan for sepsis using stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-65 years old, diagnosed with sepsis
* Clinical diagnosis of sepsis (based on Sepsis 3.0 International Guidelines)
* Confirmed or suspected infection

Exclusion Criteria:

* Violation of medical ethics
* Significant confounding factors likely to bias study outcomes
* Poor adherence to the study protocol
* Concurrent participation in other clinical trials
* Specific medical conditions:

  1. History of chronic enteritis, neuropsychiatric disorders, or transplantation (bone marrow, lung, liver, pancreas, or small intestine)
  2. Severe primary diseases affecting survival (e.g., life-limiting hepatic, renal, or endocrine disorders) or psychiatric disorders
  3. History of hypersensitivity or severe adverse reactions to biological products
  4. Imminent terminal status (e.g., septic shock, life expectancy <7 days)
  5. Foreseeable risk of medical errors or disputes during hospitalization
  6. Active drug-resistant infections
  7. History of malignancy at screening
  8. Pregnancy, lactation, or plans for pregnancy within the next year

Ages: 0 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day survival rate | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] He X, Ai S, Guo W, Yang Y, Wang Z, Jiang D, Xu X. Umbilical cord-derived mesenchymal stem (stromal) cells for treatment of severe sepsis: aphase 1 clinical trial. Transl Res. 2018 Sep;199:52-61. doi: 10.1016/j.trsl.2018.04.006. Epub 2018 Apr 30. PMID 30044959
- [Background] Li Z, Song Y, Yuan P, Guo W, Hu X, Xing W, Ao L, Tan Y, Wu X, Ao X, He X, Jiang D, Liang H, Xu X. Antibacterial Fusion Protein BPI21/LL-37 Modification Enhances the Therapeutic Efficacy of hUC-MSCs in Sepsis. Mol Ther. 2020 Aug 5;28(8):1806-1817. doi: 10.1016/j.ymthe.2020.05.014. Epub 2020 May 15. PMID 32445625
- [Background] Nemeth K, Leelahavanichkul A, Yuen PS, Mayer B, Parmelee A, Doi K, Robey PG, Leelahavanichkul K, Koller BH, Brown JM, Hu X, Jelinek I, Star RA, Mezey E. Bone marrow stromal cells attenuate sepsis via prostaglandin E(2)-dependent reprogramming of host macrophages to increase their interleukin-10 production. Nat Med. 2009 Jan;15(1):42-9. doi: 10.1038/nm.1905. Epub 2008 Nov 21. PMID 19098906
- [Background] Yagi H, Soto-Gutierrez A, Kitagawa Y, Tilles AW, Tompkins RG, Yarmush ML. Bone marrow mesenchymal stromal cells attenuate organ injury induced by LPS and burn. Cell Transplant. 2010;19(6):823-30. doi: 10.3727/096368910X508942. Epub 2010 Jun 23. PMID 20573305
- [Background] Wannemuehler TJ, Manukyan MC, Brewster BD, Rouch J, Poynter JA, Wang Y, Meldrum DR. Advances in mesenchymal stem cell research in sepsis. J Surg Res. 2012 Mar;173(1):113-26. doi: 10.1016/j.jss.2011.09.053. Epub 2011 Oct 24. PMID 22225756
- [Background] Jin HJ, Bae YK, Kim M, Kwon SJ, Jeon HB, Choi SJ, Kim SW, Yang YS, Oh W, Chang JW. Comparative analysis of human mesenchymal stem cells from bone marrow, adipose tissue, and umbilical cord blood as sources of cell therapy. Int J Mol Sci. 2013 Sep 3;14(9):17986-8001. doi: 10.3390/ijms140917986. PMID 24005862
- [Background] Yi T, Song SU. Immunomodulatory properties of mesenchymal stem cells and their therapeutic applications. Arch Pharm Res. 2012 Feb;35(2):213-21. doi: 10.1007/s12272-012-0202-z. Epub 2012 Feb 28. PMID 22370776
- [Background] Akiyama K, Chen C, Wang D, Xu X, Qu C, Yamaza T, Cai T, Chen W, Sun L, Shi S. Mesenchymal-stem-cell-induced immunoregulation involves FAS-ligand-/FAS-mediated T cell apoptosis. Cell Stem Cell. 2012 May 4;10(5):544-55. doi: 10.1016/j.stem.2012.03.007. Epub 2012 Apr 26. PMID 22542159
- [Background] Gangji V, Hauzeur JP. Cellular-based therapy for osteonecrosis. Orthop Clin North Am. 2009 Apr;40(2):213-21. doi: 10.1016/j.ocl.2008.10.009. PMID 19358906
- [Background] Phinney DG, Di Giuseppe M, Njah J, Sala E, Shiva S, St Croix CM, Stolz DB, Watkins SC, Di YP, Leikauf GD, Kolls J, Riches DW, Deiuliis G, Kaminski N, Boregowda SV, McKenna DH, Ortiz LA. Mesenchymal stem cells use extracellular vesicles to outsource mitophagy and shuttle microRNAs. Nat Commun. 2015 Oct 7;6:8472. doi: 10.1038/ncomms9472. PMID 26442449
- [Background] Kaya S. Adventure of recombinant human activated protein C in sepsis and new treatment hopes on the horizon. Recent Pat Inflamm Allergy Drug Discov. 2012 May;6(2):159-64. doi: 10.2174/187221312800166822. PMID 22292553
- [Background] Wiessner WH, Casey LC, Zbilut JP. Treatment of sepsis and septic shock: a review. Heart Lung. 1995 Sep-Oct;24(5):380-92; quiz 392-3. doi: 10.1016/s0147-9563(05)80059-7. PMID 8567303
- [Background] Fry DE. Sepsis, systemic inflammatory response, and multiple organ dysfunction: the mystery continues. Am Surg. 2012 Jan;78(1):1-8. PMID 22273282